CLINICAL TRIAL: NCT06379724
Title: The Use of Topical Tranexamic Acid Versus Thrombin Spray for the Management of Split Thickness Skin Graft Recipient Site in Burn Management
Brief Title: Burn Study- Tranexamic Acid Versus Thrombin in Split Thickness Skin Graft
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Dhaval Bhavsar, Associate Professor, Plastic, Burn and Wound Surgery, Director of Research, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 150349
Record Dates: First submitted 2023-08-21; First posted 2024-04-23 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-08

CONDITIONS: Burns; Skin Graft Complications
MeSH Terms: conditions — Burns | interventions — Tranexamic Acid; Thrombin; Skin Transplantation; Transplantation, Autologous

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, blinded, non-inferiority study
Who Masked: Participant
Masking Description: Subjects will be blinded to their randomization group. Study subject number will be linked to their randomization group. Blinding may be broken if the subject experiences an adverse reaction to the medication utilized for their group so that they are aware that they cannot receive the medication in the future. The research coordinator will have the code to the blind. The surgical team will not be blinded as the overall consistency of the topical agents will differ and may be apparent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (Active Comparator): Prior to application of the skin graft, a thin layer of thrombin is sprayed onto the wound base. The skin graft is then applied to the recipient site and fixated in standard fashion.
  Interventions: Drug: Thrombin JMI; Procedure: skin graft
- Experimental (Experimental): Tranexamic acid solution will be sprayed onto the wound base after excision and prior to skin graft appliance in the same manner as the thrombin spray in the control group
  Interventions: Drug: Tranexamic acid; Procedure: skin graft

INTERVENTIONS:
Drug: Tranexamic acid — 100mg/mL 10mL vials x2 of injectable tranexamic acid will be filled into a 20 milliliter syringe with a spray tip.
  Other Names: TXA
  Arms: Experimental
Drug: Thrombin JMI — The wound base is then sprayed with a film of Thrombin-JMI
  Other Names: Thrombin
  Arms: Control
Procedure: skin graft — Skin is taken from uninjured part of the participant's body and used to surgically cover a wound or injured area with skin that contains the epidermis and a portion of the dermis.
  Other Names: skin graft, STSG, autograft

SUMMARY:
Investigators hypothesize that topical tranexamic acid will have better or comparable efficacy to topical thrombin in reducing hematoma formation at the wound base. The purpose of the study is to demonstrate that topical tranexamic acid will be a non-inferior alternative medication to the current standard of care,THROMBIN-JMI® , and at a lower cost to the health system.

DETAILED DESCRIPTION:
1. Enrolled subjects will be randomized to the control group or the tranexamic acid experimental group. Informed consent for study participation will be obtained by a team member preoperatively and informed consent for split thickness autografting will be obtained by a surgical team member. All questions will be answered and risk/benefits/alternatives will be explained in detail to the study subject. The subject will then be taken back to the operating room and anesthesia will be induced. The surgical timeout will occur verifying subject name, medical record number, planned operation, and surgical site. The subject will be prepped and draped in a sterile manner.
2. For the control group: The recipient burn site will be excised to healthy, bleeding tissue. The wound base is then sprayed with a film of THROMBIN-JMI® and covered with telfa and pressure applied for 10 minutes to achieve hemostasis while the skin graft is being harvested. The donor site will be marked to determine the size of the autograft. Tumescent solution with a local anesthetic and epinephrine is injected with a cannula and a split thickness skin graft will be taken at 1/12 inch using a Zimmer dermatome. Prior to application of the skin graft, a thin layer of thrombin is sprayed onto the wound base. The skin graft is then applied to the recipient site and fixated in standard fashion. The donor site and recipient site were dressed according to the preference of the attending physician. The patient will then awaken from anesthesia. This procedure will typically take between 60 to 120 minutes.
3. For the experimental groups: For the first phase of the study, the procedure described above was identical to that performed to the control group with the following exceptions: 100 milligram/milliliter, 10 milliliter vials x2 of injectable tranexamic acid will be filled into a 20 milliliter syringe with a spray tip. The tranexamic acid solution will be sprayed onto the wound base after excision and prior to skin graft appliance in the same manner as the thrombin spray in the control group.
4. Post-operatively, subjects will recover from anesthesia and continue routine post-operative care in the burn unit. The first assessment will occur at 48-72 hours after surgery at the first dressing change. Dressings will be changed by the nurse or burn technician who are all well-trained and experienced in burn wound care. Assessment will require documentation of hematoma occurrence, percent graft loss by measuring dimensions of non-adherent graft, and need for reoperation. If the graft is well adherent and the patient does not have barriers to discharge, the patient will be discharged and will return to clinic for follow up at post-operative day 7-10, and at 14 days. A second and third assessment will occur at this time by either the clinic medical provider or study team member. If the patient remains inpatient, the second and third assessment will be made in the hospital.

As part of the study, an objective measured hematoma rate and percent graft take will be measured rather than estimated at the 48-72 hours, 7-10 day, and 14 day follow up period which is the current protocol for this patient population.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking
* Flame or scald burn injury
* <=10% total body surface area (TBSA) partial thickness
* <= 5% total body surface area (TBSA) deep partial or full thickness
* Skin graft harvested at 1/12 inch depth, meshed 1:1 or pie crusted if the area is a small functional area

Exclusion Criteria:

* >10% total body surface area (TBSA) partial thickness burn
* >5% total body surface area (TBSA )surgical area of burn injury (deep partial or full thickness injury)
* Traumatic or chemical burn mechanism
* Patients on immunosuppression
* Uncontrolled diabetes
* Known diagnosis of peripheral vascular disease or diagnosis at time of injury
* Pregnant women
* Patients with acquired defective color vision
* Patients with subarachnoid hemorrhage
* Patients with active intravascular clotting or known hypersensitivity reactions to tranexamic acid
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The number of participants with hematoma occurrence | Post-operative day fourteen, plus or minus two days
  dichotomous endpoint
The rate of percentage of graft take adherence amongst participants | Post-operative day fourteen, plus or minus two days
  continous endpoint
Comparison of number of participants that require re-operation | Post-operative day fourteen, plus or minus two days
  dichotomous endpoint

SECONDARY OUTCOMES:
Difference in cost between two hemostatic agents | during surgery
  The cost comparison between two hemostatic agents

CONTACTS AND LOCATIONS:
Overall Officials: Dhaval Bhavsar, MBBS, Principal Investigator — University of Kansas Medical Center
Locations (1):
- The University of Kansas Health System, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No